CLINICAL TRIAL: NCT00742196
Title: Retinal Nerve Fiber Layer Thickness Measurement on Parapapillary Atrophy With
Brief Title: Retinal Nerve Fiber Layer Thickness Measurement on Parapapillary Atrophy With the Cirrus High-Definition (HD) Optical Coherence Tomography (OCT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Gong Je Seong, Yonsei University College of Medicine
Other Study IDs: 3-2008-0076-2
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma
Keywords: Parapapillary atrophy; Retinal nerve fiber layer thickness; Glaucoma; Cirrus OCT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: No parapapillary atrophy
- 2: Parapapillary atrophy

SUMMARY:
Retinal nerve fiber layer (RNFL) thickness measurement on the parapapillary atrophy is incorrect. Because a new spectral domain OCT, the Cirrus HD OCT, uses a movable circle to analyze the RNFL thickness, we may suggest a new analysis strategy for the parapapillary atrophy.

DETAILED DESCRIPTION:
Recently, the retinal nerve fiber layer (RNFL) thickness measurement using the optical coherence tomography (OCT) becomes very useful to detect such a glaucomatous damage. However, there are some difficult cases including parapapillary atrophy to perform this measurement. Because the RNFL thickness is so sensitive to the position of measurement and the measurement of RNFL thickness on parapapillary atrophy is incorrect, it is difficult to determine exact RNFL thickness in patients with a large parapapillary atrophy. In the present study, we want to find the proper method to analyze the RNFL thickness on parapapillary atrophy. The previous OCT used a fixed circle to measure the RNFL thickness, but the new spectral domain OCT, the Cirrus HD OCT, uses a movable one. Therefore, we may suggest a new analysis strategy for the parapapillary atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Qualified OCT images (signal strength > or = 8)

Exclusion Criteria:

* Previous intraocular surgery history
* Media opacity
* DM

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with or without parapapillary atrophy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-12 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness | when the OCT images are taking
Size of parapapillary atrophy | when the OCT images are taking

CONTACTS AND LOCATIONS:
Overall Officials: Gong Je Seong, MD, PhD, Principal Investigator — Yonsei University
Locations (1):
- Gong Je Seong, Seoul, South Korea